CLINICAL TRIAL: NCT04701307
Title: Niraparib (PARP Inhibitor) Plus Dostarlimab (Anti-PD1) for Small Cell Lung Cancer (SCLC) and Other High-Grade Neuroendocrine Carcinomas (NEC)
Brief Title: Niraparib and Dostarlimab for the Treatment of Small Cell Lung Cancer and Other High-Grade Neuroendocrine Carcinomas
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0412; NCI-2020-13698 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0412 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-01-06; First posted 2021-01-08 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Lung Small Cell Carcinoma; Neuroendocrine Carcinoma; Stage III Lung Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8; Stage IIIB Lung Cancer AJCC v8; Stage IIIC Lung Cancer AJCC v8
MeSH Terms: conditions — Small Cell Lung Carcinoma; Carcinoma, Neuroendocrine; Lung Neoplasms | interventions — dostarlimab; Immunoglobulin G; Disulfides; niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (niraparib, dostarlimab) (Experimental): Patients receive niraparib PO QD on days 1-21 of cycles 1-4, and on days 1-42 of subsequent cycles. Patients also receive dostarlimab IV over 30 minutes on day 1. Cycles repeat every 21 days for cycles 1-4 and every 42 days for subsequent cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Dostarlimab; Drug: Niraparib

INTERVENTIONS:
Biological: Dostarlimab — Given IV
  Other Names: ANB011; Immunoglobulin G4, Anti-programmed Cell Death Protein 1 (PDCD1) (Humanized Clone ABT1 Gamma4-chain), Disulfide with Humanized Clone ABT1 Kappa-chain, Dimer; TSR 042; TSR-042; TSR042
Drug: Niraparib — Given PO
  Other Names: MK-4827; MK4827

SUMMARY:
This phase II trial studies the effect of niraparib and dostarlimab in treating small cell lung cancer and other high-grade neuroendocrine carcinomas. Niraparib is an inhibitor of PARP, an enzyme that helps repair deoxyribonucleic acid (DNA) when it becomes damaged. Blocking PARP may help keep cancer cells from repairing their damaged DNA, causing them to die. PARP inhibitors are a type of targeted therapy. Immunotherapy with monoclonal antibodies, such as dostarlimab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving niraparib and dostarlimab may help to control the diseases.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine objective response rate (ORR) and 6-month progression free survival (PFS) in response to combined niraparib plus dostarlimab in patients with recurrent small cell lung cancer (SCLC) and high-grade neuroendocrine carcinomas (NECs).

SECONDARY OBJECTIVES:

I. To evaluate toxicity of combined niraparib plus dostarlimab (PARP inhibition plus anti-PD-1) in patients with recurrent SCLC and other high-grade NECs.

II. To determine overall survival (OS), PFS, disease control rate (response plus stable disease > 12 weeks) to combined niraparib plus dostarlimab in patients with recurrent SCLC and other high-grade NECs.

EXPLORATORY OBJECTIVE:

I. To determine treatment-related changes in immune profiles or other biomarker in response to combined niraparib plus dostarlimab in patients with recurrent SCLC and other high-grade NECs.

OUTLINE:

Patients receive niraparib orally (PO) once daily (QD) on days 1-21 of cycles 1-4, and on days 1-42 of subsequent cycles. Patients also receive dostarlimab intravenously (IV) over 30 minutes on day 1. Cycles repeat every 21 days for cycles 1-4 and every 42 days for subsequent cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up within 90 days, every 6 months for 2 years, then annually for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have unresected or locally advanced small cell lung cancer (Cohort 1) or high-grade neuroendocrine carcinoma (Cohort 2) confirmed by staff pathologist. High-grade neuroendocrine carcinoma of prostate (e.g. aggressive variant prostate cancer, small cell of prostate, etc.) are excluded
* Patients must have had at least one prior line of systemic therapy directed at their malignancy
* Participant must have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 1
* Participant must be >= 18 years of age
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 100,000/uL
* Hemoglobin >= 9 g/dL
* Serum creatinine =< 1.5 x upper limit of normal (ULN) or calculated creatinine clearance >= 60 mL/min using the Cockcroft-Gault equation
* Total bilirubin =< 1.5 x ULN (=< 2.0 in patients with known Gilberts syndrome) OR direct bilirubin =< 1 x ULN
* Aspartate aminotransferase and alanine aminotransferase =< 2.5 x ULN unless liver metastases are present, in which case they must be =< 5 x ULN
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 x ULN unless patient is receiving anticoagulant therapy as long as PT or partial thromboplastin (PTT) is within therapeutic range of intended use of anticoagulants. Activated partial thromboplastin time (aPTT) =< 1.5 x ULN unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Participant receiving corticosteroids may continue as long as their dose equivalent to 10 mg prednisone or less and is stable for least 4 weeks prior to initiating protocol therapy
* Participant must agree to not donate blood during the study or for 90 days after the last dose of study treatment
* Female participant has a negative serum pregnancy test within 7 days prior to taking study treatment if of childbearing potential and agrees use an adequate method of contraception from screening through 180 days after the last dose of study treatment, or is of nonchildbearing potential. Nonchildbearing potential is defined as follows (by other than medical reasons):

  * >= 45 years of age and has not had menses for > 1 year
  * Patients who have been amenorrhoeic for < 2 years without history of a hysterectomy and oophorectomy must have a follicle stimulating hormone value in the postmenopausal range upon screening evaluation
  * Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure, otherwise the patient must be willing to use an adequate barrier method throughout the study, starting with the screening visit through 180 days after the last dose of study treatment. Information must be captured appropriately within the site's source documents. Note: Abstinence is acceptable if this is the established and preferred contraception for the patient
  * Pelvic irradiation
* Participant must agree to not breastfeed during the study or for 180 days after the last dose of study treatment
* Male participant agrees to use an adequate method of contraception starting with the first dose of study treatment through 180 days after the last dose of study treatment. Note: Abstinence is acceptable if this is the established and preferred contraception for the patient
* Participant must be able to understand the study procedures and agree to participate in the study by providing written informed consent
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial

Exclusion Criteria:

* Participant must not be simultaneously enrolled in any interventional clinical trial
* Participant must not have previously received a simultaneous combination of PARP inhibitor and immune checkpoint blockade (immunotherapy)
* Participant must not have had major surgery =< 3 weeks prior to initiating protocol therapy and participant must have recovered from any surgical effects
* Participant must not have received investigational therapy =< 4 weeks prior initiating protocol therapy
* Participant has had radiation therapy encompassing > 20% of the bone marrow within 2 weeks; or any radiation therapy within 1 week prior to day 1 of protocol therapy
* Participant must not have a known hypersensitivity to niraparib and dostarlimab components or excipients
* Participant must not have received a transfusion (platelets or red blood cells) =< 4 weeks prior to initiating protocol therapy
* Participant must not have received colony-stimulating factors (e.g., granulocyte colony-stimulating factor, granulocyte macrophage colony-stimulating factor, or recombinant erythropoietin) within 4 weeks prior initiating protocol therapy
* Participant has had any known grade 3 or 4 anemia, neutropenia or thrombocytopenia due to prior chemotherapy that persisted > 4 weeks and was related to the most recent treatment
* Participant must not have any known history of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML)
* Participant must not have a serious, uncontrolled medical disorder, nonmalignant systemic disease, or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 90 days) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, or any psychiatric disorder that prohibits obtaining informed consent
* Participant must not have had diagnosis, detection, or treatment of another type of cancer =< 2 years prior to initiating protocol therapy (except basal or squamous cell carcinoma of the skin and cervical cancer that has been definitively treated)
* Participant must not have known, symptomatic brain or leptomeningeal metastases. Patients should have magnetic resonance imaging (MRI) brain with and without contrast (or computed tomography [CT] head with and without contrast) within 4 weeks prior to initiation of therapy. If history of known brain metastases, these must be treated with completion of treatment at least two weeks prior to initiation of therapy. Known brain metastases must be clinically stable and asymptomatic
* Patient experienced >= grade 3 immune-related adverse event (AE) with prior immunotherapy
* Participant has a diagnosis of immunodeficiency or has received systemic steroid therapy in excess of 10 mg prednisone (or equivalent) or any other form of immunosuppressive therapy within 7 days prior to initiating protocol therapy
* Participant has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [qualitative] is detected)
* Participant has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Participant must not have a history of interstitial lung disease
* Participant has received a live vaccine within 14 days of initiating protocol therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
6-month Progression free survival (PFS) | Time from the start of study treatment to the earlier date of assessment of progression or death by any cause in the absence of progression, assessed at 6 months
  Defined as the number (or fraction) of patients who are alive without evidence of progression at 6 months from initiation of therapy. Progression will be assessed by Response Evaluation Criteria in Solid Tumors (RECIST) version (v.)1.1 criteria using investigator's review. As there is no comparator arm, the rates will be considered in the context of historical controls. Will be performed using Kaplan-Meier methods for each cohort. Quartiles (i.e. 25th percentile, median, 75th percentile) and associated two-sided 95% confidence intervals will be provided. Estimates of PFS at 6-months will be estimated from Kaplan-Meier survival curve.
Objective response rate (ORR) | At 3 months
  Defined as the percentage of patients with complete response (CR) or partial response (PR), as assessed by RECIST v.1.1 criteria using independent central review by MD Anderson Quantitative Imaging Analysis Core. As there is no comparator arm, the rates will be considered in the context of historical controls.

SECONDARY OUTCOMES:
12-week disease control rate | At 12 weeks
  Defined as the percentage of patients with CR, PR, or stable disease, as assessed by RECIST v.1.1 criteria using (independent central or investigator's) review at 12 weeks from initiation of therapy.
Progression free survival | Time from the start of study treatment to the earlier date of assessment of progression or death by any cause in the absence of progression, assessed up to 12 months
  Progression will be assessed by RECIST v.1.1 criteria using investigator's review. Will be performed using Kaplan-Meier methods for each cohort. Quartiles (i.e. 25th percentile, median, 75th percentile) and associated two-sided 95% confidence intervals will be provided. Estimates of PFS at 6-months and 12-months will be estimated from Kaplan-Meier survival curve.
Overall survival (OS) | From the start of study treatment to the date of death by any cause, assessed up to 5 years
  Will be performed using Kaplan-Meier methods for each cohort. Quartiles (i.e. 25th percentile, median, 75th percentile) and associated two-sided 95% confidence intervals will be provided. Estimates of OS at 6-months and 12-months will be estimated from Kaplan-Meier survival curve.
Incidence of adverse events (AEs) | Up to 90 days post-treatment
  Defined as frequency and grade of adverse events. All AEs will be assessed by the investigator for severity according to Common Terminology Criteria for Adverse Events v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Carl M Gay, MD,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MDAndersonCancerCenterWebsite — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2021-08-05): https://cdn.clinicaltrials.gov/large-docs/07/NCT04701307/ICF_000.pdf